CLINICAL TRIAL: NCT02962271
Title: Comparation of Ultrasonic Imaging of Enthesopathy in Patients With Psoriatic Arthritis and Psoriasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhu, Clinical Professor, Chinese PLA General Hospital
Other Study IDs: ChinaPLAGH-PsA
Record Dates: First submitted 2016-11-03; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Enthesopathy
Keywords: Musculoskeletal Ultrasound; Psoriatic Arthritis; Enthesopathy
MeSH Terms: conditions — Enthesopathy; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Psoriatic Arthritis: Musculoskeletal ultrasound (MSUS) of the lower limbs' entheses were performed
  Interventions: Device: Musculoskeletal Ultrasound
- Psoriasis: Musculoskeletal ultrasound (MSUS) of the lower limbs' entheses were performed
  Interventions: Device: Musculoskeletal Ultrasound

INTERVENTIONS:
Device: Musculoskeletal Ultrasound — Musculoskeletal ultrasound (MSUS) of the lower limbs' entheses were performed

SUMMARY:
Psoriatic arthritis(PsA) and psoriasis(Ps) are two systemic inflammatory diseases linked with rash of psoriasis, but there's still great controversy regarding the exact relationship between them. Our study is to investigate the characteristics and differences of the ultrasonic imaging of enthesopathy in the lower extremity in patients with PsA and Ps, to explore the risk factors of Ps developing into PsA in the long term course.

DETAILED DESCRIPTION:
As one of the most common chronic inflammatory skin diseases, psoriasis(Ps) can be intimately associated to psoriatic arthritis (PsA), affecting approximately 1% to 2% of the world's population. About 30% of them will develop into PsA with serious impact on their health-related quality of life.

PsA, characterised by different subsets with varying degree of severity, is a chronic, complicated inflammatory disease.Enthesitis is the prevalent and distinctive feature of PsA.

Musculoskeletal Ultrasound (MSUS) is a valid noninvasive modality, essential to evaluate entheses thickness, enthesophytes, bursitis and bone erosions as well as to disclose vascularisation on tendons through power doppler (PD) assessment. In recent years, more and more attention has been paid to the diagnosis and management of Ps and PsA, owing to its discrimination of identifying subclinical entheses and joint changes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of plaque psoriasis, psoriatic arthritis, ankylosing spondylitis, rheumatoid arthritis or osteoarthritis.
* Body Mass Index (BMI)<30 kg/m2.
* Absence of local glucocorticoid or other drugs injection or surgical treatment for entheses scanned in the previous 6 weeks prior to clinical and musculoskeletal ultrasound (MSUS) evaluation.

Exclusion Criteria:

* Other systemic rheumatic diseases or malignant neoplasms.
* Peripheral neuropathy of lower extremity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A series of 44 patients with PsA, 44 age- and sex-matched patients of Ps and 44 HCs consecutively admitted from the outpatients clinic and ward from January 2016 to September 2016.
Sampling Method: Probability Sample
Enrollment: 187 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The rate of enthesopathy comparison between psoriatic arthritis(PsA) and psoriasis(Ps) as assessed by SPSS v17.0 | up to 10 months

SECONDARY OUTCOMES:
The potential risk factors of Ps for PsA as assessed by SPSS v17.0 | up to 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhu, Principal Investigator — Department of Rheumatology,PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) are to be shared with other researchers, whenever it will be available, and it may be obtained by requesting from the principal investigator